CLINICAL TRIAL: NCT01051934
Title: A Phase I Trial of SS1 (dsFv) PE38 With Paclitaxel, Carboplatin, and Bevacizumab in Subjects With Unresectable Non-Small Cell Lung Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100032; 10-C-0032; NCT01041118 (obsolete NCT alias)
Record Dates: First submitted 2010-01-16; First posted 2010-01-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-09-28

CONDITIONS: Non-Small Cell Lung Cancer; Adenocarcinoma
Keywords: Recombinant Immunotoxin; Monoclonal Antibody; Pseudomonas Exotoxin; Targeted Therapy; Lung Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Lung Neoplasms | interventions — SS1(dsFv)PE38; Paclitaxel; Carboplatin; Bevacizumab

INTERVENTIONS:
Drug: SS1 (dsFv) PE38
Drug: Paclitaxel
Drug: Carboplatin
Drug: Bevacizumab

SUMMARY:
Background:

* Advanced cases of non-small-cell lung carcinoma (NSCLC) usually are not successfully treated with standard therapies. Even treatments that attempt to specifically target NSCLC cells have not proved effective.
* Researchers are interested in determining whether a combination of the chemotherapy drugs SS1 (dsFv) PE38, paclitaxel, carboplatin, and bevacizumab may be effective in shrinking the size of NSCLC tumors. Three of the drugs (paclitaxel, carboplatin, and bevacizumab) are commercially available, while the other is a drug that is currently being tested to determine its usefulness in cancer treatment. This study will help to determine if the combination of all four drugs is more effective and as safe, safer, or less safe than other drug combinations given to treat NSCLC.

Objectives:

- To determine a safe and tolerable dose for the combination of SS1 (dsFv) PE38 with paclitaxel, carboplatin, and bevacizumab in patients with advanced mesothelin-expressing lung adenocarcinoma.

Eligibility:

* Age > 18 years of age
* Newly diagnosed advanced non-small-cell lung carcinoma
* No prior chemotherapy for lung cancer
* Individuals at least 18 years of age who have advanced non-small-cell lung carcinoma that has not responded to standard treatments.

Design:

* The study will last for two 21-day cycles of treatment for the four-drug combination, with additional treatment cycles of carboplatin, paclitaxel, and bevacizumab.
* Two to three weeks prior to the study, participants will be screened with a full medical history and physical exam, bone marrow biopsy (we do not do bone marrow biopsies) (if one has not been performed in the last 6 months), computed tomography (CT) or ultrasound scan, tumor measurements, and other tests as required by the researchers. Participants will provide blood and urine samples at this time as well.
* During the study, participants will receive SS1 (dsFv) PE38, carboplatin, paclitaxel, and bevacizumab for a maximum of two cycles. On Day 15 of the first cycle, participants will provide a blood sample to be tested to see if SS1 (dsFv) PE38 is being effective. If the tests show that SS1 (dsFv) PE38 is not effective, participants will not receive another dose of it, but will continue to receive paclitaxel, carboplatin, and bevacizumab for the second cycle.
* After the first two cycles, participants will continue to receive carboplatin, paclitaxel, and bevacizumab every 3 weeks for up t...

DETAILED DESCRIPTION:
* Treatment with platinum-based doublet chemotherapy results in a median survival of 7 to 10 months in patients with locally advanced or metastatic non-small cell lung cancer.
* In a randomized clinical trial of patients with non-squamous cell lung cancer, treatment with carboplatin, paclitaxel and bevacizumab resulted in an objective response rate of 35%, overall survival of 12.3 months compared to objective response rate of 15%, overall survival of 10.3 months in patients treated with carboplatin and paclitaxel alone.
* Mesothelin is a cell surface glycoprotein present on normal mesothelial cells that is highly expressed in many human cancers including lung adenocarcinoma.
* SS1 (dsFv) PE38 is a recombinant anti-mesothelin immunotoxin that has undergone phase I testing and is currently in clinical trials in combination with pemetrexed and cisplatin for treatment of malignant pleural mesothelioma.
* Pre-clinical studies demonstrate increased anti-tumor activity of SS1 (dsFv) PE38 in combination with chemotherapy and bevacizumab against mesothelin-expressing tumors.

Primary Objectives:

- This is a phase I study to determine a safe and tolerable phase II dose for the combination of SS1 (dsFv) PE38 with paclitaxel, carboplatin and bevacizumab in patients with advanced mesothelin-expressing lung adenocarcinoma.

Secondary Objectives:

* To assess response rate, duration of response, and progression-free survival (PFS).
* To characterize the pharmacokinetics (PK) of SS1 (dsFv) PE38 in combination with chemotherapy and bevacizumab.
* Monitor serum mesothelin levels prior to and during chemotherapy.
* To identify T-cell epitopes responsible for neutralizing SS1 (dsFv) PE38 activity using mononuclear cells obtained by apheresis.

Eligibility:

* Histologically confirmed stage IIIB (malignant pleural effusion) or IV or recurrent NSCLC (non-squamous cell, with mesothelin expression greater than or equal to 10% of tumor cells by IHC).
* Adequate organ and bone marrow function.
* ECOG performance status of 0-1.

Design:

- Open label phase I trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Histologically or cytologically documented non-small cell lung adenocarcinoma that is confirmed by the Laboratory of Pathology, NIH.
  2. Mesothelin expression greater than or equal to 10% of tumor cells as determined by immunohistochemistry (IHC) on tumor tissue specimens.
  3. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral CT scan.
  4. Stage IIIB (malignant pleural effusion) or stage IV non-small cell lung cancer or recurrent non-small cell lung cancer.
  5. Age greater than or equal to 18 years (males or non-pregnant females).
  6. Life expectancy of greater than 3 months.
  7. ECOG performance status 0-1 (Karnofsky > 60%).
  8. Serum Creatinine less than or equal to 1.5mg/dl.
  9. Hemoglobin greater than or equal to 10.0g/dl.
  10. Absolute neutrophil count greater than or equal to 1,500/m(3) and platelets greater than or equal to 100,000/m(3).
  11. AST/SGOT and ALT/SGPT less than or equal to 2.5 times ULN, total bilirubin less than or equal to 1.5 times ULN (In patients with evidence of Gilberts disease, elevated bilirubin should not be related to tumor or other liver diseases and should be less than or equal 2 times upper limit of normal).
  12. Urine protein to creatinine ratio < 1.0.
  13. The ability to understand and the willingness to sign a written informed consent document and the ability to comply with the requirements of the protocol. The effects of SS1 (dsFv) PE38 on the developing human fetus are unknown. For this reason and because immunotoxins are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for at least 3 months thereafter. Women of childbearing potential must have a negative pregnancy at study enrollment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Inclusion of Women and Minorities:

Both men and women and members of all races and ethnic groups are eligible for this trial.

EXCLUSION CRITERIA:

1. Squamous cell cancer or mixed tumors with any small cell element.
2. Tumor of any histology in close proximity to a major vessel or cavitation.
3. History of hemoptysis (bright red blood of teaspoon or more (greater than or equal to 2.5 mL)) on one occasion unrelated to any diagnostic procedure within the past year.
4. Patients with CNS metastases.
5. History of uncontrolled hypertension, defined as blood pressure > 140/90 mmHg (NCI CTEP Active Version of the CTCAE grade greater than or equal to 2) are excluded. However, these patients will be eligible if the blood pressure is < 140/90 mmHg after anti-hypertensive treatment.
6. Any of the following within 6 months prior to study enrollment: myocardial infarction, unstable angina pectoris or uncontrolled angina pectoris, coronary/peripheral artery bypass graft, NYHA class III or IV congestive heart failure, clinically significant peripheral vascular disease (Grade II or greater). History of stroke or transient ischemic attack within 6 months.
7. Psychiatric or neurologic illness that would limit compliance with study requirements.
8. Patients with serious illness or medical condition.
9. Severe active infection within 14 days requiring use of intravenous antibiotics before beginning treatment.
10. Patients may not be receiving any other investigational agents.
11. History of an active malignancy unless curatively treated and risk of recurrence of < 5% at five years other than in situ carcinoma of the cervix, or non-melanomatous skin cancers.
12. Patients must not be on therapeutic anticoagulation, chronic daily treatment with aspirin 325mg/day or non steroidal anti-inflammatory agents, or any agent known to inhibit platelet function, within 10 days prior to day 1 on study. Low dose aspirin 81mg/day is allowed.
13. History of pulmonary embolism, deep venous thrombosis or other thromboembolic event within 6 months.
14. Patients with a history of severe hypersensitivity reaction to compounds of similar chemical or biologic composition to carboplatin, paclitaxel, bevacizumab or other agents used in the study.
15. History of a major surgical procedure, open biopsy, or a significant traumatic injury within 35 days prior to commencing treatment, or the anticipation of the need for a major surgical procedure during the course of the study prior to the predetermined date of tumor excision. Fine needle aspirations or core biopsies within 7 days prior to commencing treatment are allowed.
16. History of abdominal fistula, gastrointestinal perforation, intra- abdominal abscess or tracheo-esophageal fistula.
17. Non-healing wound or ulcer.
18. Evidence of coagulopathic disorder or hemorrhagic diathesis. INR greater than 1.5.
19. Pregnancy (positive pregnancy test) or active breast feeding.
20. Urine protein: creatinine ratio greater than or equal to 1.0 at screening.
21. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with chemotherapy. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
22. Significant laboratory abnormality requiring further investigation that may cause undue risk for the subject's safety, inhibit protocol participation, or interfere with interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-12-29; Primary Completion 2011-09-28 (Actual); Study Completion 2011-09-28 (Actual)

PRIMARY OUTCOMES:
Determined safe and tolerable phase 2 dose for combination of SS1 (dsFv) PE38 with paclitaxel, carboplatin, and bevacizumab.

SECONDARY OUTCOMES:
Study pharmacokinetics. Assess response rate, duration of response and progression-free survival.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chang K, Pastan I. Molecular cloning of mesothelin, a differentiation antigen present on mesothelium, mesotheliomas, and ovarian cancers. Proc Natl Acad Sci U S A. 1996 Jan 9;93(1):136-40. doi: 10.1073/pnas.93.1.136. PMID 8552591
- [Background] Folkman J. Tumor angiogenesis: therapeutic implications. N Engl J Med. 1971 Nov 18;285(21):1182-6. doi: 10.1056/NEJM197111182852108. No abstract available. PMID 4938153
- [Background] Hassan R, Bera T, Pastan I. Mesothelin: a new target for immunotherapy. Clin Cancer Res. 2004 Jun 15;10(12 Pt 1):3937-42. doi: 10.1158/1078-0432.CCR-03-0801. PMID 15217923